CLINICAL TRIAL: NCT05712577
Title: Psychological Help in Patients With Marfan Syndrome: the Role of Quality of Life, Coping Mechanisms, Psychosocial Aspects and Self-esteem Levels
Brief Title: Psychological Support in Adult Patients With Marfan Syndrome
Acronym: MARFANPSY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Alessandro Pini, Principal Investigator, IRCCS Policlinico S. Donato
Other Study IDs: MarfanPsy
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Rare Diseases; Marfan Syndrome; Psychology, Social
Keywords: Marfan syndrome; Psychological support; Self-report
MeSH Terms: conditions — Rare Diseases; Marfan Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MFS_PT+: MFS patients who followed psychological support/psychotherapy
  Interventions: Other: Questionnaire
- MFS_PT-: MFS patients who never followed psychological support/psychotherapy
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Rosenberg Self- Esteem scale
Other: Questionnaire — Short Form 36 scale
Other: Questionnaire — Coping orientation to the problems experienced - New Version in Italian
Other: Questionnaire — Outcome Questionnaire - version 42.5

SUMMARY:
The goal of this observational study is to identify key factors leading to psychotherapy or psychological support in adult subjects with Marfan syndrome (MSF). the main questions it aims to answer are:

* Understand and define which internal variables of the individual drive this request for psychological support;
* To learn about verify the impact that the clinical manifestations of MSF have on psychosocial aspects, self-esteem, subjective perception of the disease and coping mechanisms.

DETAILED DESCRIPTION:
Patients following psychological interview during follow-up visits will be enrolled in the study.

The following self-report questionnaires will be used in understanding the impact the syndrome has on mental health and quality of life:

* Rosenberg Self- Esteem: 10 item Likert scale for assessing self-esteem;
* SF 36: 36 item scale assessing eight domains: physical functioning physical role limitations; bodily pain; general health perceptions; energy/vitality; social functioning; emotional role limitations and mental health;
* Cope NVI: to test measures coping behaviors as potential responses to stressors like social support, avoidance strategies, positive attitude, problem orientation and transcendent orientation;
* OQ45.2: measure of general psychological distress.

ELIGIBILITY:
Inclusion Criteria:

* Subjects affected by Marfan syndrome;
* Subjects currently in follow-up at Cardiovascular Genetic Centre, IRCCS Policlinico San Donato;
* Signed informed consent.

Exclusion Criteria:

* Subjects with cognitive deficits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with MFS who have requested psychological support/psychotherapy and patients who have never requested psychological support/psychotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-10-09 (Estimated); Study Completion 2024-10-09 (Estimated)

PRIMARY OUTCOMES:
Questionnaire performance | 8 Months
  Statistical analysis between the two experimental groups using independent samples t-tests for continuous variables and associations for categorical variables.
  Questionnaire scoring:
  - COPE NVI: scoring between 60 and 240; higher score means better outcome
Questionnaire performance | 8 Months
  Statistical analysis between the two experimental groups using independent samples t-tests for continuous variables and associations for categorical variables.
  Questionnaire scoring:
  - Short Form-36: scoring between 0 and 100; higher score means better outcome
Questionnaire performance | 8 Months
  Statistical analysis between the two experimental groups using independent samples t-tests for continuous variables and associations for categorical variables.
  Questionnaire scoring:
  - Rosenberg Self- Esteem scale: scoring between 0 and 30; higher score means better outcome
Questionnaire performance | 8 Months
  Statistical analysis between the two experimental groups using independent samples t-tests for continuous variables and associations for categorical variables.
  Questionnaire scoring:
  - Outcome questionnaire 42.5: socring between 0 and 180; clinical cut-off value is 64, higher score means worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Pini, MD, Principal Investigator — Cardiovascular-Gentic Centre, IRCCS Policlinico San Donato
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Lombardy, Italy